CLINICAL TRIAL: NCT05899517
Title: The Effects of Orally Administered Oxytocin on Behavioral and Neural Responses to Self Versus Other Touch Distinction
Brief Title: Oxytocin Effects on Self Versus Other Touch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-92
Record Dates: First submitted 2023-05-05; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Oxytocin; Affective touch; Self versus other distinction; fMRI
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind within-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral oxytocin then placebo (Experimental): Subjects will first receive oral lollipop with oxytocin (24IU). After a washout period of 2 weeks, they will then receive oral lollipop with placebo (identical ingredients, except the active agent).
  Interventions: Drug: oral lollipop with oxytocin (24IU); Drug: oral lollipop with placebo
- Oral placebo then oxytocin (Experimental): Subjects will first receive oral lollipop with placebo (identical ingredients, except the active agent). After a washout period of 2 weeks, they will then receive oral lollipop with oxytocin (24 IU).
  Interventions: Drug: oral lollipop with oxytocin (24IU); Drug: oral lollipop with placebo

INTERVENTIONS:
Drug: oral lollipop with oxytocin (24IU) — For oral oxytocin administration, participants will be instructed to suck the lollipop medicated with 24IU oxytocin for 3 minutes and then to sit relaxed in a quiet room for 30 minutes prior to rate their mood (PANAS). Participants then start the self versus other touch task around 53 minutes after oxytocin administration.
  Other Names: oral oxytocin
Drug: oral lollipop with placebo — For placebo administration, participants will be instructed to suck the placebo lollipop for 3 minutes and then to sit relaxed in a quiet room for 30 minutes prior to rate their mood (PANAS). Participants then start the self versus other touch task around 53 minutes after placebo administration.
  Other Names: oral placebo

SUMMARY:
The main aim of the study is to investigate the modulatory effects of oxytocin (24IU) administered orally using medicated lollipops on the behavioral and neural responses to touching yourself compared with being touched by others.

DETAILED DESCRIPTION:
In a double-blind placebo-controlled within-subject experimental design, 40 adult male subjects will be randomly allocated to either receive oral oxytocin (24IU, medicated lollipop) or placebo (lollipop without oxytocin). Starting 45 minutes after treatment a resting state functional magnetic resonance imaging (fMRI) will be recorded (8min) and next subjects will be applied two different types of stroking touch (self- vs. other-produced touch) to their left arm repeated in 16 blocks. After each block of applied touch stimulation, subjects will be required to rate their perceived pleasantness of touch from -4 (extremely unpleasant) to 4 (extremely pleasant). The neural basis of touch processing will be measured via simultaneously acquired fMRI.

To control potential confounding effects among subjects, before the experiment all participants will be asked to complete a range of Chinese versions of validated questionnaires on personality, traits, attitude towards interpersonal touch and interoceptive ability: Autism Spectrum Quotient (ASQ), Beck Depression Inventory II (BDI), State-Trait Anxiety Inventory (STAI), Social Touch Questionnaire (STQ),Sensory Over-Responsivity (SensOR) Scales, Interpersonal Reactivity Index (C-IRI), Self-Concept Clarity Scale (SCCS), Interoceptive Confusion Questionnaire(ICQ) and Multidimensional Assessment of Interoceptive Awareness(MAIA) scale. Additionally, to control for potential confounding effects of treatment on mood across the experiment, the Positive and Negative Affect Schedule (PANAS) will be administered immediately before and 30 minutes after the treatment. Participants will also complete the PANAS after the touch stimulations to further measure the modulatory effects of touch on mood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders and without any current psychotherapeutic medication.

Exclusion Criteria:

* Any history of brain injury, psychiatric/physical illness, alcohol/substance abuse, or other major health concern.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Neural index: fMRI based measures of altered neural activity in response to different types of applied touch | 53-75 minutes after treatment administration
  fMRI-based indices of neural activation (blood oxygen level dependent changes) in response to repeated self vs other touch will be compared between subjects in the oxytocin and placebo administration groups.
Behavioral index: pleasantness ratings for the different types of applied touch | 53-75 minutes after treatment administration
  Ratings of perceived pleasantness for the two types of repeatedly applied touch (after each block of touch, subjects will need to complete the question 'how pleasant do they feel for the applied touch?' using a 9-point Likert scale ranging from -4 to +4, with higher positive scores indicating greater perceived pleasantness and higher negative scores indicating greater unpleasantness) will be compared between the oxytocin and placebo administration groups.

SECONDARY OUTCOMES:
Questionnaire scores for autistic traits using the Autism Spectrum Quotient (ASQ) | Before the experiment
  Mean and standard deviation of the Autism Spectrum Quotient (ASQ) scores (0~50, higher scores mean higher autistic trait) will be computed as a measurement of autistic traits.
Questionnaire scores for attitudes towards touch using the Social Touch Questionnaire | Before the experiment
  Mean and standard deviation of the Social Touch Questionnaire (STQ) scores (0~80, higher scores mean higher aversion to touch) will be computed to measure individual attitudes towards social touch of daily life.
Questionnaire scores for self-concept using the Self-Concept Clarity Scale (SCCS) | Before the experiment
  Mean and standard deviation of the Self-Concept Clarity Scale (SCCS) scores (0~60, higher scores mean clearer self-concept) will be computed to measure clarity level of one's self-concept.
Behavioral associations with autistic traits using the Autism Spectrum Quotient (ASQ) | Before the experiment
  Associations between the Autism Spectrum Quotient (ASQ) scores (0~50, higher scores mean higher autistic trait) with behavioral rating scores (-4 to +4, with higher positive scores indicating greater perceived pleasantness and higher negative scores indicating greater unpleasantness) will be calculated to investigate modulatory effects of autistic traits.
Neural associations with autistic traits using the Autism Spectrum Quotient (ASQ) | Before the experiment
  Associations between the Autism Spectrum Quotient (ASQ) scores (0~50, higher scores mean higher autistic trait) with fMRI-based indices of neural activation (blood oxygen level dependent changes) will be calculated to investigate modulatory effects of autistic traits.
Behavioral associations with questionnaire scores for attitudes towards touch using the Social Touch Questionnaire Questionnaire (STQ) | Before the experiment
  Associations between the Social Touch Questionnaire (STQ) scores (0~80, higher scores mean higher aversion to touch) with behavioral rating scores (-4 to +4, with higher positive scores indicating greater perceived pleasantness and higher negative scores indicating greater unpleasantness) will be calculated to investigate modulatory effects of how much subjects like being touched.
Neural associations with questionnaire scores for attitudes towards touch using the Social Touch Questionnaire (STQ) | Before the experiment
  Associations between the Social Touch Questionnaire (STQ) scores (0~80, higher scores mean higher aversion to touch) with fMRI-based indices of neural activation (blood oxygen level dependent changes) will be calculated to investigate modulatory effects of how much subjects like being touched.
Behavioral associations with questionnaire scores for self-concept using the Self-Concept Clarity Scale (SCCS) | Before the experiment
  Associations between the Self-Concept Clarity Scale (SCCS) scores (0~60, higher scores mean clearer self-concept) with behavioral rating scores (-4 to +4, with higher positive scores indicating greater perceived pleasantness and higher negative scores indicating greater unpleasantness) will be calculated to investigate modulatory effects of self-concept.
Neural associations with questionnaire scores for self-concept using the Self-Concept Clarity Scale (SCCS) | Before the experiment
  Associations between the Self-Concept Clarity Scale (SCCS) scores (0~60, higher scores mean clearer self-concept) with fMRI-based indices of neural activation (blood oxygen level dependent changes) will be calculated to investigate modulatory effects of self-concept.
Resting state fMRI connectivity | 45-53 minutes after treatment
  The effects of oxytocin on resting state functional connectivity will be analyzed by comparing the strength of functional connections between pairs of regions using time-series signal measures (-1 to +1 with greater positive values indicating stronger functional connectivity) in subjects in the oxytocin and placebo treatment groups.
Resting state fMRI connectivity association with behavioral responses to touch | 45-53 minutes after treatment for resting state and 53-75 minutes after treatment for behavioral measures
  Associations between resting state fMRI connectivity and primary outcome measures will be calculated to investigate whether resting state functional connectivity is predictive of observed treatment effects on individual behavioral responses (behavioral rating scores: -4 to +4, with higher positive scores indicating greater perceived pleasantness and higher negative scores indicating greater unpleasantness) to touch.
Resting state fMRI connectivity and questionnaire scores of Autism Spectrum Quotient (ASQ) for measuring autistic traits | Pre-treatment for ASQ and 45-53 minutes after treatment for resting state
  Associations between resting state fMRI connectivity and Autism Spectrum Quotient (ASQ) scores (0~50, higher scores mean higher autistic trait) will be calculated to investigate whether resting state functional connectivity is predictive of individual autistic traits.
Resting state fMRI connectivity and questionnaire scores of Social Touch Questionnaire (STQ) for measuring responses to touch | Pre-treatment for STQ and 45-53 minutes after treatment for resting state
  Associations between resting state fMRI connectivity and Social Touch Questionnaire (STQ) scores (0~80, higher scores mean higher aversion to touch) will be calculated to investigate whether resting state functional connectivity is predictive of how much subjects like being touched.
Resting state fMRI connectivity and questionnaire scores of Self-Concept Clarity Scale (SCCS) for measuring self-concept | Pre-treatment for SCCS and 45-53 minutes after treatment for resting state
  Associations between resting state fMRI connectivity and Self-Concept Clarity Scale (SCCS) scores (0~60, higher scores mean clearer self-concept) will be calculated to investigate whether resting state functional connectivity is predictive of self-concept.

CONTACTS AND LOCATIONS:
Overall Officials: Siying Wang, Dr., Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Sichuan, China